CLINICAL TRIAL: NCT03825783
Title: Gene Therapy for Leukocyte Adhesion Deficiency-I (LAD-I): A Phase I Clinical Trial to Evaluate the Safety and Efficacy of the Infusion of Autologous Hematopoietic Stem Cells Transduced With a Lentiviral Vector Encoding the ITGB2 Gene.
Brief Title: A Gene Therapy Trial to Evaluate the Safety and Efficacy of RP-L201 in Subjects With Leukocyte Adhesion Deficiency-I
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients were enrolled under global Phase 1/2 protocol RP-L201-0318.
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L201-0218
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Leukocyte Adhesion Defect - Type I
Keywords: Leukocyte Adhesion Deficiency- Type I; LAD-I
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RP-L201 (Experimental): RP-L201 is a gene therapy product containing autologous genetically modified CD34+ hematopoietic stem cells transduced with Chim-CD18-WPRE lentiviral vector administered as a single infusion in subjects with severe LAD-I
  Interventions: Biological: RP-L201

INTERVENTIONS:
Biological: RP-L201 — CD34+ enriched hematopoietic stem cells from subjects with severe LAD-I transduced ex vivo with lentiviral vector carrying the ITGB2 gene, Chim-CD18-WPRE.

SUMMARY:
The primary purpose of the Phase I portion of the study is to determine the safety profile and preliminary evidence of efficacy associated with infusion of autologous gene-corrected hematopoietic stem cells.

DETAILED DESCRIPTION:
The study is a pediatric non-randomized open-label Phase I clinical trial. This will include a safety evaluation and preliminary assessment of the efficacy of hematopoietic gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the ITGB2 gene in subjects with severe Leukocyte Adhesion Deficiency-I (LAD-I). Subjects will undergo mobilization and collection of peripheral blood hematopoietic stem cells (HSCs) with granulocyte-colony stimulating factor (G-CSF) and plerixafor or bone marrow harvest in select circumstances.

HSCs will then be transduced with the therapeutic vector (Chim.hCD18-LV), with the intent of enabling stable integration of the provirus in the genome of stem and progenitor cells.

If the number of CD34+ cells that are cryopreserved is at least 4×10E6 total CD34+ cells/kg, subjects will receive myeloablative conditioning with intravenous busulfan. The gene-modified CD34+ cells will be then transplanted back into the subject.

Once engrafted, it is anticipated that the gene-modified stem and progenitor cells will enable hematopoiesis, generating blood cells in which the integrated therapeutic gene (ITGB2) will be transcribed and translated to produce the therapeutic CD18 protein with a preferential high expression in mature myeloid cells. Leukocytes expressing a functional CD18 will have the capability to arrest on endothelial surfaces and extravasate to infectious sites, enabling a competent antimicrobial response and reversing the clinical disorder.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of severe LAD-I as demonstrated by flow cytometry indicating CD18 expression on <2% neutrophils (polymorphonuclear neutrophils [PMNs]). (Patients in which CD18+ PMNs are >2% will be considered eligible with <2% CD11a or CD11b expressing PMNs and if there is a documented ITGB2 mutation and clinical history consistent with LAD-I (or known family history).
* At least one (1) prior significant bacterial or fungal infection (US National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], v5.0, Grade ≥2). This criteria is not required for patients with documented family history who meet the above inclusion criteria.
* Age ≥3 months.
* Considered to be an appropriate candidate for autologous transplantation of HSCs.
* A competent custodial parent with legal capacity to execute an Ethics Committee (EC)-approved consent form must be available to participate in the consent process. (Informed assent will be sought from capable patients, in accordance with the directive of the EC and with local requirements.)
* Ability to comply with trial procedures including investigational therapy and follow-up evaluations.

Exclusion Criteria:

* Availability of a medically-eligible human leukocyte antigen (HLA)-identical sibling donor transplant. Patients may not be included in this trial as an alternative to a clinically-indicated and feasible HLA-matched sibling donor HSC transplant. If an HLA-identical sibling is identified, but mobilized peripheral blood or bone marrow HSC collection is not feasible (for example: donor is in utero, is a newborn from whom cord blood was not collected, or is unable to undergo donation procedure because of medical impairments), then inclusion may be permitted per the Principal Investigator discretion.
* Hepatic dysfunction as defined by either:

  * Bilirubin > 1.5 × the upper limit of normal (ULN) or
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5×ULN
* Pulmonary dysfunction as defined by either:

  * Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection).
  * Oxygen saturation (by pulse oximetry) <90%.
* Evidence of active metastatic or locoregionally advanced malignancy (including hematologic malignancy) for which survival is anticipated to be less than 3 years.
* Serious infections with persistent bloodstream pathogens at time of trial entry. (Patients with active infections [e.g., unresolved ulcerative lesions, skin or oral infections] are permitted as long as appropriate antibiotic therapy has been [or is being] administered).
* Any medical or other contraindication for both leukopheresis and bone marrow harvest procedure, as determined by the treating investigator.
* Any medical or other contraindication for the administration of conditioning therapy, as determined by the treating investigator.
* Significant medical conditions, including documented human immunodeficiency virus (HIV) infection, poorly-controlled diabetes, poorly-controlled hypertension, poorly-controlled cardiac arrhythmia or congestive heart failure; or arterial thromboembolic events (including stroke or myocardial infarction) within the 6 prior months.
* Any medical or psychiatric condition that in the opinion of the Principal Investigator renders the patient unfit for trial participation or at higher than acceptable risk for participation.

Patients who are evaluated for the trial and determined ineligible may be subsequently evaluated and declared eligible if the criteria by which they were considered ineligible is reversible (for example: bloodstream infection, transient increase in liver enzymes) and there is documented and plausible evidence of its resolution in the opinion of the Principal Investigator.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by United States (US) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 | 2 years
  Evaluation of safety associated with treatment with RP-L201
Survival following infusion of RP-L201 | 2 years
  Evaluation of survival as determined by the proportion of subjects alive at age 2 (24 months) and at least 1-year post infusion without allogeneic hematopoietic stem cell transplant

SECONDARY OUTCOMES:
CD18 expression after infusion of RP-L201 | 2 years
  Determination of the percentage of subjects in whom infusion of RP-L201 results in a change in the percentage of neutrophils expressing CD18 to at least 10% in 2 years
Genetic correction after infusion of RP-L201 | 6 months
  Determination of whether infusion of RP-L201 results in vector copy number/cell of at least 0.1 in peripheral blood neutrophils carrying the therapeutic Chim.hCD18-LV provirus at 6 months post-infusion
Incidence of infections after infusion of RP-L201 | 2 years
  Determination of the incidence and severity of bacterial or other infections (subsequent to hematopoietic reconstitution)
Assessment of number of participants with a change in LAD-I-associated neutrophilia after infusion of RP-L201 | 2 years
  Evaluation of change to partially normal or to normal levels of LAD-I-associated neutrophilia
Assessment of number of participants with a change in skin lesions or periodontal abnormalities after infusion of RP-L201 | 2 years
  Evaluation of resolution (partial or complete) of any underlying skin lesions or periodontal abnormalities
Assessment of overall survival after infusion of RP-L201 | 2 years
  Evaluation of overall survival (beyond age 2 years and beyond the initial year subsequent to investigational therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Julián Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús (HIUNJ)
Locations (1):
- Hospital Infantil Universitario Niño Jesús (HIUNJ), Madrid, Spain